CLINICAL TRIAL: NCT05364060
Title: Assessment of Severe Depression Related to Psychotrauma in the COVID-19 Context in Patients Followed in Psychiatry in the Department of Eure
Brief Title: COVID-19 and Mental Health in Eure
Acronym: COVID-SME
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Eure-Seine (Other)
Collaborators: New Hospital of Navarre (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2021-A01280-41; CHES N°21/02 (Other: CH Eure-Seine)
Record Dates: First submitted 2022-05-05; First posted 2022-05-06 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: COVID-19 Pandemic; Psychiatric Disorder
Keywords: covid-19; psychiatry
MeSH Terms: conditions — COVID-19; Mental Disorders | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients followed in psychiatry: Quantitative questionnaires
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — Different questionnaires detailed in the objectives part

SUMMARY:
Research Hypothesis: Living conditions during COVID-19, and lockdowns and curfews impact the psychological state of patients (assessed by the degree of depression, positive and negative thoughts, insomnia, state of post-traumatic stress).

DETAILED DESCRIPTION:
From the early stages of the COVID-19 pandemic, concerns were raised about its effect on mental health and on patients with mental illness. Several surveys and cross-sectional assessments, in Italy, England, Ecuador and China in 2020, have suggested that patients with COVID-19 have symptoms of anxiety (including stress disorder traumatic, depression and insomnia.

In France, a survey by "Santé Publique France" on the impact of COVID-19 on mental health carried out in November 2020, revealed a 20% rate of depressive symptoms in the general population.

The objective of this study is to assess the level of psychological distress and the prevalence of psychiatric disorders related to COVID-19 as part of the follow-up of psychiatric patients in the department of Eure since March 2020, which has coincided with the onset of the health crisis, including consecutive lockdowns and curfews.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Coming for a psychiatric consultation or hospitalization at the New Hospital of Navarre or in the extra-hospital centers of the department of Eure
* Patient who has received the information note and who does not refuse to participate in the study

Exclusion Criteria:

* Patient not understanding French
* Patient followed in psychiatry for a major cognitive disorder
* Patient under legal protection measure (guardianship, curatorship, safeguard of justice, future protection mandate or family authorization)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients coming for a psychiatric consultation or hospitalization at the New Hospital of Navarre or in the extra-hospital centers of the department of Eure
Sampling Method: Probability Sample
Enrollment: 585 (Estimated)
Dates: Start 2022-06-13 (Actual); Primary Completion 2023-06-13 (Estimated); Study Completion 2023-06-13 (Estimated)

PRIMARY OUTCOMES:
Evaluation of prevalence of severe depression in patients followed in psychiatry in the department of Eure | Baseline
  The scale used is BDI-FS-Fr (Beck Depression Inventory-Fast Screen-French) scale, composed of seven self-assessment items taken from the 21 items of the BDI-II. The BDI-FS-Fr has been validated in France.

SECONDARY OUTCOMES:
Describe population characteristics | Baseline
  Typical demographic information such as age, gender, education level, current living situation, etc, and characteristics related to COVID-19
Evaluation of sleep disorder | Baseline
  It will be effectuated via the Insomnia Severity Index (ISI) that is a self-reported measure assessing the subjective symptoms and consequences of insomnia, as well as the degree of worry or distress caused by sleep difficulties. The French version of the ISI has also been validated.
Evaluation of post-traumatic stress disorder | Baseline
  The evaluation of post-traumatic stress disorder is performed via the SPAN (Startle, Physiological arousal, Anger, and Numbness) scale. The SPAN is a four-item scale for post-traumatic stress disorder that was empirically derived from the DTS (Davidson Trauma Scale).
  The minimum value for this scale is 0, the maximum, 16. Higher scores mean a worse outcome.
Evaluation of positive and negative thoughts | Baseline
  Both positive and negative thoughts will be assessed using two positive and negative thought screening thermometers. Scoring is calculated from 0 to 10 for each scale.

CONTACTS AND LOCATIONS:
Overall Officials: Tarik Mazouzi, MD, Principal Investigator — New Hospital of Navarre
Locations (1):
- CH Eure-Seine, Évreux, France

IPD SHARING:
Plan to Share IPD: No